CLINICAL TRIAL: NCT05917548
Title: Development and Pilot Implementation of an Oral Health Promotion Strategy Mediated by Teledentistry Focused on Community-dwelling Older Adults of the La Araucanía Region of Chile
Brief Title: Oral Health Promotion Mediated by Teledentistry in Community-dwelling Older Adults of La Araucanía Region, Chile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fernanda Muñoz Sepúlveda (Other)
Collaborators: Subvención Presidencial, Ministerio de Hacienda, Chile (Unknown); Centro Interuniversitario de Envejecimiento Saludable (CIES) (Unknown); Beca de Postgrado Magíster Nacional, ANID (Unknown)
Responsible Party: Sponsor-Investigator, Fernanda Muñoz Sepúlveda, Principal Investigator, Universidad de La Frontera
Organization: Universidad de La Frontera (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 082/22
Record Dates: First submitted 2023-06-06; First posted 2023-06-26 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Oral Health Knowledge; Oral Health Attitudes; Oral Health Self-efficacy
Keywords: Teledentistry; Oral health promotion; Elderly

STUDY DESIGN:
Intervention Model Description: The participants were contacted via phone calls for enrolment in TEGO platform where the pre-test of knowledge, attitudes and oral health self-efficacy was applied. Then, they were scheduled for medical-dental-geriatric diagnosis in a mobile dental clinic where all receive a standardized face-to-face oral health individual education. The investigator in charge of sending the videos performed age-stratified randomization in every city of the study using a random number generator function of the Epidat 4.2 program for the allocation of the participants in comparison or intervention groups. The videos were sent to the participants in the intervention group, this information is masked for the dental care providers and for the outcome assessor. 6 weeks later the face-to-face intervention both groups were assessed in with the post-test via phone call.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The random assignment was blinded for the dental care provider, outcome assesor and for the co-investigator in charge of the statistical analysis. (Double-blind RCT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-education (Experimental): The tele-education group will receive the same intervention as the comparison group with an educational reinforcement mediated by teledentistry. This intervention consists of 4 educational videos, designed for the elderly, promoting correct toothbrushing and flossing, detection, and prevention of dental caries, periodontal disease, and oral cancer. These four videos were sent via WhatsApp.
  Interventions: Device: Teledentistry oral health promotion; Behavioral: Face-to-Face oral health promotion
- Comparison (Active Comparator): The comparison group receive a medical-dental-geriatric diagnosis and face-to-face standardized education via powerpoint presentation and use of dental models for the promotion of correct toothbrushing and flossing, detection, and prevention of dental caries, periodontal disease, and oral cancer.
  Interventions: Behavioral: Face-to-Face oral health promotion

INTERVENTIONS:
Device: Teledentistry oral health promotion — Educational videos specially designed and validated for elderly (duration 4 to 6 minutes each one)
  Arms: Tele-education
Behavioral: Face-to-Face oral health promotion — Standardized PowerPoint presentation of 15 minutes about the most common or dangerous oral diseases (dental caries, periodontal disease and oral cancer), and toothbrushing and flossing practice in dental models

SUMMARY:
The goal of this randomized clinical trial is to compare the knowledge, attitudes, and oral health self-efficacy in self-sufficient elders aged over 60 years of 4 cities of La Araucanía región, Chile.

The main questions it aims to answer are:

* Can the development and implementation of a teledentistry strategy focused on community-dwelling older adults of the La Araucanía region improve participants' knowledge, attitudes, and self-efficacy in oral health?
* Could this teledentistry strategy have acceptability greater than 80%?

Participants will receive a dental-medical-geriatric diagnosis in a mobile dental clinic supported by a web platform called Teleplatform of Geriatric Dental Specialties (TEGO) and individual oral health education.

The researchers will compare a comparison group that will receive face-to-face individual oral health education with an intervention group, called tele-education group, that will receive educational reinforcement through a teledentistry strategy mediated by oral health educational videos sent via WhatsApp; to see if there are differences in the knowledge, attitudes, and oral health self-efficacy between the groups.

DETAILED DESCRIPTION:
Access to oral health promotion for the elderly has been limited during their lifetime. The purpose of this study is the development and pilot implementation of an oral health promotion strategy mediated by teledentistry focused on community-dwelling older adults of the La Araucanía region. To this end, a randomized clinical trial is proposed with pre- and post-intervention tests to be carried out in a sample (n:120) of people over 60 years of age from 4 cities in this region. Both groups will undergo a dental-medical-geriatric diagnosis in a mobile dental clinic supported by a web platform called Teleplatform of Geriatric Dental Specialties (TEGO) and individual oral health education. The intervention group will also receive educational reinforcement through oral health videos sent via WhatsApp (Tele-education). The strategy will be evaluated through a questionnaire of knowledge, attitudes and self-efficacy in oral health that will be applied before and after the interventions received by both groups. The acceptability of the tele-educational strategy will be assessed. The statistical analysis contemplates the description of the sociodemographic profiles of the participants and the acceptability perceived by those who make up the tele-education group. The average of the scores obtained in the pre and post-test of the questionnaire will be compared within each group through the T-test for related samples and the average of the final scores will be compared between both groups through the T-test for independent samples. Likewise, the relationship between the post-test results, sociodemographic variables, and clinical variables will be evaluated through the Pearson Correlation Coefficient. A value of p < 0.05 was chosen as the threshold for significance.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 60 years of age residing in La Araucanía Region
* Self-valent (Barthel index ≥ 90)
* With access to a smartphone and internet
* Ability to follow instructions and adequate mobility to go up to a mobile dental clinic.

Exclusion Criteria:

* Subjects with cognitive impairment (Folstein Mini-Mental ≤ 24)
* Totally edentulous
* Those who do not use WhatsApp

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-10-14 (Actual)

PRIMARY OUTCOMES:
Change in oral health knowledge | Change from baseline oral health knowledges at 6 weeks
  Questionnaire of 38 items focused on identifying signs and symptoms of dental caries, periodontal disease, and oral cancer, as well as preventive measures for each condition. The responses for signs and symptoms were quantified using a 'Yes' , 'I don't know' or 'No' scale, while preventive measures were ranked on a 5-point scale ranging from 'Very important to 'Not at all important
Change in oral health attitudes | Change from baseline oral health attitudes at 6 weeks
  Attitudes were measured via a 5-point scale, which evaluated seven items associated with the inevitability of oral disease in the elderly, the value of keeping natural teeth, and the effectiveness of preventive behaviors
Change in oral health self-efficacy | Change from baseline oral health self-efficacy at 6 weeks
  Oral Health self-efficacy scale to assess the individual's confidence in their ability to prevent oral diseases. This survey has 8 items under the subordinate categories of oral and general health self-efficacy, six and two questions respectively. All of the eight items had to be rated along a five-point Likert scale comprising Not at all Confident, Not confident, Neither confident nor unconfident, Confident, and Strongly Confident ratings.

SECONDARY OUTCOMES:
Acceptability: Utility of the teledentistry intervention | 2 days after sending each video
  The utility of each video was assesed via a 4-point scale
Acceptability: Dropout rate | Change from baseline up to 6 weeks
  Percentage withdrawal of study participants
Acceptability: Recomendation | After 6 weeks
  Binary question with a yes or no answer on whether you would recommend this type of care and promotion of oral health to friends and/or family

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Dental Móvil TEGO-UFRO, Temuco, La Araucanía, Chile

IPD SHARING:
Plan to Share IPD: Yes
All IPD underlying the results will be shared in one publication
Supporting Information: Study Protocol
Time Frame: When summary data are published

REFERENCES:
- [Background] Beltran V, Flores M, Sanzana C, Munoz-Sepulveda F, Alvarado E, Venegas B, Molina JC, Rueda-Velasquez S, von Marttens A. Tooth Loss and Caries Experience of Elderly Chileans in the Context of the COVID-19 Pandemic in Five Regions of Chile. Int J Environ Res Public Health. 2023 Feb 9;20(4):3001. doi: 10.3390/ijerph20043001. PMID 36833696
- [Background] Beltran V, von Marttens A, Acuna-Mardones P, Sanzana-Luengo C, Rueda-Velasquez SJ, Alvarado E, Flores M, Cerda A, Venegas B. Implementation of a Teledentistry Platform for Dental Emergencies for the Elderly in the Context of the COVID-19 Pandemic in Chile. Biomed Res Int. 2022 Mar 22;2022:6889285. doi: 10.1155/2022/6889285. eCollection 2022. PMID 35330690